CLINICAL TRIAL: NCT02370576
Title: The Effect of Traumatic Childbirth on the Incidence of Postpartum PTSD, MDD and Anxiety Disorders
Brief Title: The Effect of Traumatic Childbirth on the Incidence of PTSD and Other Major Postpartum Psychopathology
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Marina Bar-Shai, MD, PhD, MD, PhD, Rambam Health Care Campus
Other Study IDs: rambam001
Record Dates: First submitted 2015-02-15; First posted 2015-02-25 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-02

CONDITIONS: Stress Disorders, Post-Traumatic; Depressive Disorder, Major
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- control: Healthy women after elective cesarean section.Questionnaire/ rating scale application. Screening: protocol designed to assess or examine methods of identifying a condition (or risk factors for a condition) in people who are not yet known to have the condition (or risk factor).
  Interventions: Other: rating scale application
- emergency: Healthy women after emergency cesarean section. Questionnaire/ rating scale application. Screening: protocol designed to assess or examine methods of identifying a condition (or risk factors for a condition) in people who are not yet known to have the condition (or risk factor).
  Interventions: Other: rating scale application

INTERVENTIONS:
Other: rating scale application — Administration of validated PTSD, MDD and anxiety disorders rating scales immediately after birth and 1 month postpartum.
  rating scale application
  Other Names: rating scale

SUMMARY:
Determination of incidence and prevalence of PTSD and other types of psychopathology (such as anxiety and affective disorders) after traumatic birth experiences and elucidation of salient risk factors in the local population sample- by prospective follow-up.

DETAILED DESCRIPTION:
Post- traumatic stress disorder (PTSD)- definitions The criteria for the diagnosis of traumatic experience involve the experience of a specific traumatic stressor and, subsequently, four axes of symptoms: (i) re-experiencing of the traumatic event, including nightmares, intrusive thoughts and emotions; (ii) avoidance of stimuli associated with the traumatic event; (iii) hyperarousal, expressed as difficulties sleeping or concentrating, irritability, enhanced startle responses, irritable, aggressive, reckless or self-destructive behavior and (iv) persistent negative alterations in cognitions and mood. Formal clinical diagnosis of PTSD can only be made after symptoms have been present for at least 1 month. The definition of a traumatic event includes the witnessing or experience of serious threat to life or bodily integrity, or injury (either physical or emotional) to oneself or others [1]. As such, the subjective and objective experience of giving birth became recognized as a possibly traumatic event for some women [2]. As a result of a traumatic childbirth, women may experience general distress, flashbacks, dissociation, amnesia, sleep disturbances, negative evaluation of self-worth, difficulty breastfeeding, relationship problems and problems with their own sexuality [3-7], problems with bonding with their infants [8-12], or significant fear of subsequent childbirth (tocophobia); many choose not to conceive again for this reason. The afflicted women that do choose to have further children may insist on a cesarean delivery in hopes that it will not be as traumatic [6].

PTSD after childbirth- prevalence, risk factors, clinical characteristics and long term implications About 2- 6% of women will experience the full DSM-V criteria for PTSD at some point after giving birth [13-14]. An additional 22- 40% may meet the criteria for subsyndromal PTSD, and another 20-50% of women may report the childbirth experience as traumatic [13-14].

It is not known at this point what are the characteristics of women who may develop postpartum PTSD, making it impossible to predict or to prevent this outcome. However, several risk factors have been recently elucidated. Several predisposing/prenatal factors associated with the childbirth experience itself have been associated with PTSD. These include previous psychiatric history [15, 16, 17,18] (especially depression in pregnancy), socio-demographic problems [19,20, 21] (lack of support, problematic relationship with the partner), parity (primiparous more at risk), personality traits and disorders [22 -24] (trait anxiety; anxiety sensitivity, neuroticism), previous trauma [25-26]

* previous childbirth-related trauma; sexual abuse), maladaptive cognitions [27] (pre-existing, maladaptive schemas; negative cognitive appraisal of past childbirth; autobiographical memory specificity, fear of upcoming childbirth), nature of delivery [28, 29] (type and number of interventions; duration, fear of harm to self or baby, emergency cesarean section (CS), instrumental delivery- especially forceps- assisted, episiotomy), perception of care from medical staff [24, 29], perception of loss of control [24, 30], perception of pain [24 ], infant complications [28-29] (especially low birth weight, low Apgar score, asphyxia, resuscitation, prematurity), and peritraumatic dissociation [31-32] - feeling of unreality; alterations in perception of time and place; feeling of disconnection from body). Women having unplanned caesarean section births were likely to report PTSD-type symptoms. However, there was no association between PTSD type symptoms and planned caesarean section births [16, 33]. PTSD is also associated with preeclampsia [34-35]. Preeclampsia is associated with both maternal complications (e.g. eclampsia, abruptio placentae, pulmonary edema, acute renal failure) [36-37], and perinatal complications (e.g. fetal growth restriction, preterm delivery, and perinatal death) [38, 39-40]. As previously described, these adverse pregnancy outcomes are known to be associated with PTSD [41, 43, 44 -46]. Other seemingly routine aspects of pregnancy may increase vulnerability to active PTSD, especially in victims childhood sexual trauma or intrafamilial abuse [47, 48, 3-4], previous pregnancy loss [5,6 ] or prior traumatic birth [7], or when pregnancy is a result of sexual assault. Inherent physical aspects of pregnancy such as increased breast sensitivity and fetal movement are potentially triggering. Routine aspects of prenatal care, including vaginal and breast examinations, can be triggers, especially for sexual trauma survivors. Labor itself, especially medicalised labor can exacerbate a sense of powerlessness and vulnerability, which can trigger PTSD symptoms [49]. Physical changes of pregnancy, especially cardiovascular, respiratory, gastrointestinal and renal system alterations, also could affect the experience of PTSD symptoms [49], since they might resemble physical sensations associated with anxiety.

It is unclear whether traumatic birth experiences can lead to other types of psychopathology, such as postpartum depression or anxiety disorders, and more research is needed to answer this question. However, since there is a known association between traumatic experiences and affective and anxiety disorders in general- one can surmise that this association exists also between these disorders and traumatic birth experiences [10, 12, 16].

It is now believed that PTSD severity after childbirth reaches a plateau over the 12 months postpartum, without further improvement, which means that women with postpartum PTSD do not spontaneously recover [50]. Thus, many afflicted women develop a chronic disorder that significantly interferes with their functioning in various areas of life. PTSD during the postpartum period is an important public health issue because of the longer-term negative impact of maternal mental health problems on child development [8] including impaired mother-infant relationship [9-10], delayed intellectual development [11,12 ], and psychiatric disorder in children [51]. In many PTSD patients the baby can become a constant reminder of the traumatic birth. Some women report that they felt guilty for blaming the baby after a traumatic childbirth experience. PTSD within 11 months postpartum is associated with depression within 11 months postpartum. Little is known about mother-child bonding in women with PTSD after childbirth, while the negative impact of maternal postnatal depression on child development has been investigated by different authors showing that especially chronicity of maternal depression after birth is a predictor for negative development [28, 12].

PTSD after childbirth- pathophysiology Pregnancy is associated with alterations in the hypothalamic-pituitary-ovarian (HPO) axis, particularly increases in plasma concentrations of progesterone and estrogen, which can modulate mood and cognition. Pregnancy also is associated with changes in the hypothalamic-pituitary-adrenal (HPA) axis, including increases in plasma adrenocorticotropic hormone and cortisol, and a large increase in plasma corticotropin-releasing hormone, especially in the third trimester (from placental secretion) [16].

In addition to being a stress hormone, cortisol appears to affect memory, salience, social cognition, negative mood, [52] alertness and sleep [52]. It is possible that the altered hormonal milieu of both HPA and HPO axes in pregnancy could affect the expression of PTSD symptoms by increasing frequency and emotional intensity of traumatic memories, which in turn affect mood, motivation, social cognition, sleep, and concentration [33].

PTSD after childbirth- assessment tools. Several validated rating scales are in use in PTSD research. The gold standard is Clinician-Administered PTSD Scale for DSM-5 (CAPS-5), which is rated by a researcher and necessitates time and experience in its administration. PTSD Symptoms Scale (PSS) and PTSD Checklist for DSM-5 (PCL-5) are self- report short rating scales. Also in use are depression rating scales such as Montgomery- Asberg Depression Rating Scale (MADRS, researcher- administered), Major Depression Inventory (MDI, self- report) and Edingurgh Postnatal Depression Scale (EPDS, self- report, specifically created to assess the symptoms of peri- and postpartum depression) [53].

Research goals. Determination of incidence and prevalence of PTSD and other types of psychopathology (such as anxiety and affective disorders) after traumatic birth experiences and elucidation of salient risk factors in the local population sample- by prospective follow-up.

Materials and methods We shall apply to the local Helsinki Committee to receive the approval for the research. The participants will receive an explanation and sign informed consent.

Compare a cohort of women with perinatal complications (emergency CS, instrumental deliveries, premature labor, serious hemorrhage at childbirth, perineal tear that required stitching, resuscitation of the newborn, newborn admitted to neonatal intensive care unit) to a control cohort of healthy women who delivered by elective uncomplicated CS. For women in both cohorts it should be their first pregnancy and first childbirth. Assess with the help of rating scales (both researcher- administered and self- report, such as CAPS, PCL-C, MADRS, MDI, EPDS) in the first two days following childbirth to measure the baseline parameters and to assess the prevalence of acute stress reaction (ASR) in the research and the control cohorts. Assess again both cohorts by the above methods 1 month after childbirth. Compare the prevalence of PTSD between the different cohorts of perinatal complications and the control cohort. Also- compare the prevalence of PTSD, anxiety and mood disorders between the different groups of perinatal complications in order to determine which type of complication carries the greater risk for the development of psychopathology. Determine whether the development of ASR 2 days after childbirth is predictive of PTSD and other types of psychopathology 1 month after childbirth. Thus- determine the prevalence of PTSD and other types of psychopathology 1 month after birth in risk groups versus controls, prospectively.

ELIGIBILITY:
Inclusion Criteria:

* No psychiatric background

Exclusion Criteria:

* Known psychiatric disorder

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Either healthy women without previous psychiatric background,1-2 days after an uncomplicated planned Cesarean birth, or healthy women without previous psychiatric background, 1-2 days after an emergency Cesarean birth.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of PTSD (Questionnaire/ rating scale application) | 1 month

SECONDARY OUTCOMES:
Presence or absence of major depression (Questionnaire/ rating scale application) | 1 month
Presence or absence of anxiety disorders (Questionnaire/ rating scale application) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Marina Bar-Shai, MD, PhD, Principal Investigator — Rambam Healthcare Center
Locations (1):
- Rambam Medical Center, Haifa, Israel